CLINICAL TRIAL: NCT02822222
Title: A Phase 1/2, Randomized, Double-Blind, Placebo-Controlled Study to Assess the Safety and Tolerability of RMJH-111b in Adult Subjects With Essential Hypertension
Brief Title: Safety Study of RMJH-111b to Treat Essential Hypertension
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: RMJ Holdings, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: RMJH-111b-002
Record Dates: First submitted 2016-06-28; First posted 2016-07-04 (Estimated); Results first posted 2020-09-23 (Actual); Last update posted 2020-09-23 (Actual); Status verified 2020-09

CONDITIONS: Essential Hypertension
Keywords: essential hypertension; hypertension; high blood pressure; cardiovascular disease; RMJH-111b; magnesium; magnesium citrate; calcium channel blocker; vasodilator; antihypertensive; anti-hypertensive
MeSH Terms: conditions — Essential Hypertension; Hypertension; Cardiovascular Diseases | interventions — magnesium citrate

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: This study was a double-blind, placebo-controlled study. The Investigational Site pharmacist was not blinded and was responsible for dispensing the appropriate study drug based upon the randomization schedule and ensuring that the remaining Investigational Site personnel were blinded to the drug.
  Total serum magnesium was used to monitor for magnesium toxicity and subjects with levels ≥ 5 mg/dL were to be discontinued. Thus, there was the potential for these measurements to unblind the Principal Investigator. Due to the pre-existing endogenous levels of total serum magnesium and urine magnesium and the relatively large variability in values between subjects, review of these numbers would not necessarily have suggested one treatment arm over the other. To minimize the impact of such potential unblinding on the ABPM endpoints, a centralized ABPM reader was used and the reader was blinded to the total serum magnesium and urine magnesium values.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- RMJH-111b (Experimental): Four (4) RMJH-111b (magnesium citrate, tribasic anhydrous) soft gelatin capsules (110 mg elemental magnesium/capsule) orally bid for 7 days
  Interventions: Drug: Magnesium citrate, tribasic anhydrous soft gelatin capsule
- Placebo (Placebo Comparator): Four (4) placebo soft gelatin capsules (0 mg elemental magnesium/capsule) orally bid for 7 days
  Interventions: Drug: Placebo soft gelatin capsule

INTERVENTIONS:
Drug: Magnesium citrate, tribasic anhydrous soft gelatin capsule — 110 mg elemental magnesium/capsule
  Other Names: RMJH-111b
  Arms: RMJH-111b
Drug: Placebo soft gelatin capsule — 0 mg elemental magnesium/capsule
  Other Names: Placebo
  Arms: Placebo

SUMMARY:
The purpose of this study was to evaluate the safety of RMJH-111b, including how well it is tolerated, and the effect of RMJH-111b on blood pressure in subjects with hypertension. The study also measured the amount of magnesium in the blood and urine before and after RMJH-111b administration to evaluate what the body does to RMJH-111b (pharmacokinetics).

DETAILED DESCRIPTION:
This was a phase 1/2, single center, randomized, double-blind, placebo-controlled study to assess the safety and tolerability of RMJH-111b in adult subjects with essential hypertension. Assessments of pharmacokinetics and efficacy were secondary objectives.

RMJ Holdings LLC (doing business as RMJH Rx) is developing RMJH-111b (magnesium citrate, tribasic anhydrous) soft gelatin capsules for the treatment of essential hypertension. The rationale for developing RMJH-111b for essential hypertension is based on reported calcium channel blocker and vasodilator effects of magnesium cation (Mg++). Given this hypothesized mechanism of action, RMJH-111b may not be effective for subjects with other causes or forms of hypertension, and thus the diagnosis of essential hypertension was a key inclusion criterion for this trial.

In order to avoid confounding the results of the trial, subjects who were already taking anti-hypertensive medications to manage their hypertension were taken off of those medications and underwent a 7-day washout period. Subjects that met the specified blood pressure criteria after the washout [systolic blood pressure (SBP) ≥ 150 and ≤ 200 mmHg and diastolic blood pressure (DBP) ≥ 95 and ≤ 115 mmHg] received placebo orally twice a day (bid) for a 3-day run-in period (Days 1-3). Subjects that were recently diagnosed or previously diagnosed and off treatment for > 1 week before starting the study and who met the blood pressure criteria proceeded directly to the 3-day run-in period (i.e., without the 7-day washout period). During the 3-day run-in period, the subjects remained in the clinical research unit (CRU) on a low salt (2.5 g/24 hours) diet.

Subjects that remained eligible after the run-in period were randomized to receive either 440 mg of RMJH-111b or placebo orally bid (i.e., total daily dose of 880 and 0 mg elemental magnesium, respectively) for a 7-day treatment period (Days 4-10). A total of 21 subjects randomized 15:6 to RMJH-111b or placebo was planned. Subjects were randomized on either June 10th or 23rd of 2016. Based on the screen failure rate of the 1st cohort, the number of subjects needed for the 2nd cohort was projected. The actual number of subjects eligible for randomization at the end of the run-in period in the 2nd cohort exceeded the projection by 1 and all eligible subjects were randomized. Thus, the actual number of subjects randomized was 22, with 16 subjects in the RMJH-111b group and 6 subjects in the placebo group (i.e., 16:6 rather than 15:6). Subjects remained in the CRU on a low salt (2.5 g/24 hours) diet for the entire 7-day treatment period and through the 24-hour post treatment assessments (Day 11).

Subjects returned to the clinic 8 days (±3 days) after the last dose of Study Drug (active or placebo) for their Final Study Visit.

Protocol-specified reasons for discontinuing a subject from the study included, but were not limited to: 1) subject's blood pressure was too elevated for them to safely continue in the study (subjects who experienced SBP >200 mmHg or DBP >115 mmHg had to have these measurements repeated approximately 1 hour later, and if the SBP or DBP remained elevated, the subject was to be removed from the study and treated accordingly), 2) subject experienced a sharp drop in blood pressure (SBP < 110 mmHg or DBP < 60 mmHg); 3) subject's patellar reflex (knee jerk) disappeared, and 4) subject's total serum magnesium levels increased to ≥ 5 mg/dL (twice the upper limit of normal). As a conservative measure for this first trial of RMJH-111b, the criterion regarding drop in blood pressure did not require any associated clinical symptoms. For the pivotal trial, RMJH Rx will incorporate orthostatic hypotension monitoring and refine the discontinuation criterion regarding drop in blood pressure to allow for continued Study Drug treatment in the absence of clinical symptoms, so as to avoid unnecessarily removing a subject that is experiencing therapeutic benefit.

All measurements used for the safety assessments in this study are widely used, and generally recognized as reliable, accurate, and relevant. Further, they included standard parameters used in the evaluation of drugs with the potential for anti-hypertensive and magnesium toxicity effects.

Because blood pressure varies at daytime compared to nighttime, mean daytime (8 AM to 4 PM), nighttime (10 PM to 6 AM), and 24-hour ambulatory blood pressure monitor (ABPM) parameters were used to assess the efficacy effects of RMJH-111b on blood pressure in this trial. While 24-hour ambulatory blood pressure monitoring is considered as a more precise method for the evaluation of drug effects on blood pressure than clinic visit (seated) blood pressures, this trial also included efficacy evaluations of seated SBP and DBP parameters for informational purposes and in particular to facilitate the design of the larger pivotal trial where ABPM monitoring will not be practical.

The pharmacokinetic (PK) evaluation of magnesium is complicated by pre-existing endogenous levels of magnesium, other ingested sources of magnesium (daily diet and supplements; supplements with total daily dose of magnesium ≤ 150 mg were allowed in this study), and the tight regulation of magnesium in the body (magnesium homeostasis) with relatively high levels of magnesium in bones and soft tissues compared to approximately 1% in the blood. Thus, the total serum magnesium exposure was anticipated to be minimally effected with RMJH-111b intake, but evidence of urinary magnesium excretion coupled with maintained total serum magnesium exposure was expected to provide an indication of intake rather than magnesium wasting.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, 18-80 years old
* Diagnosed with essential hypertension
* SBP ≥ 150 & ≤ 200 mmHg & DBP ≥ 95 and ≤ 115 mmHg after resting for 5 minutes in the seated position at Day 1 & baseline (pre-dose Day 4)
* Both males & women of child bearing potential (WCBP) agree to use adequate contraceptive methods while on study
* Willing and able to sign informed consent form (ICF)
* Suitable for participation in the study in the opinion of the Investigator

Exclusion Criteria:

* History of myocardial infarction, congestive heart failure, or stroke within 6 months of Screening, or evidence of greater than 1st degree heart block or myocardial damage
* History of chronic hepatitis
* Uncontrolled diabetes (hemoglobin A1C ≥ 6.5%) at Screening or Day 1
* Glomerular filtration rate < 60 mL/min at Screening or Day 1
* Serum hypo- or hyper-natremia (≤ 133 & ≥145 meq/L) at Screening or Day 1
* Low serum potassium (≤ 3.3 meq/L) at Screening or Day 1
* Low total serum magnesium (≤ 1.3 mg/dL) or total serum magnesium greater than the upper limit of normal (2.5 mg/dL) at Screening or Day 1
* Serum uric acid > 6.5 mg/dL for females or >7.5 mg/dL for males at Screening or Day 1
* Absence of patellar reflex (knee jerk) at Day 1-3, or pre-dose Day 4
* Evidence of clinically significant findings at Screening, during the run-in period (Days 1-3), or at baseline (pre-dose Day 4) which, in the opinion of the Investigator would pose a safety risk or interfere with appropriate interpretation of safety data
* Malignancy within 5 years of the Screening Visit (with the exception of basal cell and squamous cell skin carcinoma)
* Major surgery within four weeks prior to Screening
* Presence of a malabsorption syndrome possibly affecting drug absorption (e.g., Crohn's disease or chronic pancreatitis)
* Presence of irritable bowel syndrome, ulcerative colitis, or chronic diarrhea
* History of psychotic disorder
* History of alcoholism or drug addiction or current alcohol or drug use that, in the opinion of the Investigator, will interfere with the subject's ability to comply with the dosing schedule & study evaluations
* History of any illicit drug use within one year prior to Screening
* Positive drug screen at Screening or at Day 1, except subjects on prescription drugs that in the opinion of the Investigator will not influence the outcome of the study
* Positive breathalyzer test for blood alcohol content at Screening or at Day 1
* Consumption of more than five cups of caffeinated beverages per day
* Current treatment or treatment within 30 days prior to the first dose of Study Drug (active or placebo; Day 4) with another investigational drug, or current enrollment in another clinical trial
* Current treatment or treatment within 10 days prior to the first dose of Study Drug (active or placebo; Day 4) with any anti-hypertension medication (other than Study Drug during the treatment period)
* Current treatment or treatment within 30 days prior to the first dose of Study Drug (active or placebo; Day 4) with magnesium-containing antacids or laxatives, dietary supplement(s) where the total daily dose of magnesium is greater than 150 mg, central nervous system depressants, neuromuscular blocking agents, or cardiac glycosides, lithium-containing drugs, bisphosphonates, sodium polystyrene sulfonate, or tetracycline/quinolone antibiotics, anti-tumor necrosis factor-alpha drugs, or phytotherapeutic/herbal/ plant derived preparations
* Known hypersensitivity to magnesium
* Known hypersensitivity to the inactive ingredients in the Study Drug (placebo and active)
* Positive pregnancy test at Screening or at Day 1, or lactating
* Arm circumference greater than 42 centimeters

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2016-06-10 (Actual); Primary Completion 2016-07-07 (Actual); Study Completion 2016-07-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joel M Neutel, MD, Principal Investigator — Orange County Research Center
Locations (1):
- Orange County Research Center, Tustin, California, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This trial was conducted at a single Investigational Site (Orange County Research Center) in Tustin, CA. All subject recruitment procedures and materials were reviewed & approved by a central IRB prior to their use. The 1st screening visit was May 31, 2016, the 1st subject was enrolled on June 10, 2016, & the last subject visit was July 7, 2016.
Pre-assignment Details: Randomization to treatment took place on Day 4, following the 7-day washout period & the 3-day run-in placebo period. Only subjects that continued to meet eligibility criteria following the Day 4 baseline procedures were randomized.
Period: Overall Study
Arm/Group | RMJH-111b | Placebo
Started (Number started means number randomized to treatment at Day 4.) | 16 | 6
Completed | 15 | 6
Not Completed | 1 | 0
Not completed — Protocol requirement SBP<110 mmHg | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | RMJH-111b | Placebo | Total
Number analyzed (Participants) | 16 | 6 | 22
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 14 | 4 | 18
  >=65 years | 2 | 2 | 4
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.08 (8.882) | 61.36 (5.889) | 58.98 (8.175)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 0 | 8
  Male | 8 | 6 | 14
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 1 | 2
  Not Hispanic or Latino | 15 | 5 | 20
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 1
  Black or African American | 9 | 3 | 12
  White | 5 | 3 | 8
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 16 | 6 | 22
Height [Mean (Standard Deviation); unit: cm] — Baseline height was measured at the Screening visit using a calibrated stadiometer with the subject wearing no shoes.
  cm | 170.3 (8.79) | 174.0 (10.43) | 171.3 (9.16)
Weight [Mean (Standard Deviation); unit: kg] — Baseline weight was measured after the washout period and before the first placebo run-in dose (i.e., on Day 1) using a calibrated scale with the subject wearing light clothes and no shoes.
  kg | 90.54 (14.865) | 89.35 (9.492) | 90.21 (13.401)
Heart rate [Mean (Standard Deviation); unit: beats per minute] — Baseline heart rate was measured after the run-in period and prior to the first randomized dose (i.e., pre-dose Day 4). The measurement was made after the subject was sitting for at least 5 minutes in a quiet environment and prior to the blood sample collection for baseline total serum magnesium.
  beats per minute | 72.50 (7.572) | 66.33 (8.710) | 70.82 (8.180)
Respiration rate [Mean (Standard Deviation); unit: breaths per minute] — Baseline respiration rate was measured after the run-in period and prior to the first randomized dose (i.e., pre-dose Day 4). The measurement was made after the subject was sitting for at least 5 minutes in a quiet environment and prior to the blood sample collection for baseline total serum magnesium.
  breaths per minute | 12.75 (1.000) | 12.33 (0.816) | 12.64 (0.953)
Temperature [Mean (Standard Deviation); unit: degrees Celsius] — Baseline temperature was measured after the run-in period and prior to the first randomized dose (i.e., pre-dose Day 4).
  degrees Celsius | 36.59 (0.208) | 36.60 (0.063) | 36.60 (0.179)
Seated SBP [Mean (Standard Deviation); unit: mmHg] — Baseline seated SBP was measured after the run-in period and prior to the first randomized dose (i.e., pre-dose Day 4). The measurement was made after the subject was sitting for at least 5 minutes in a quiet environment and prior to the blood sample collection for baseline total serum magnesium. The recorded seated SBP value was the mean of two measurements taken 2 minutes apart and using the dominant arm.
  mmHg | 160.4 (8.58) | 162.0 (5.06) | 160.9 (7.69)
Seated DBP [Mean (Standard Deviation); unit: mmHg] — Baseline seated DBP was measured after the run-in period and prior to the first randomized dose (i.e., pre-dose Day 4). The measurement was made after the subject was sitting for at least 5 minutes in a quiet environment and prior to the blood sample collection for baseline total serum magnesium. The recorded seated DBP value was the mean of two measurements taken 2 minutes apart and using the dominant arm.
  mmHg | 101.4 (5.18) | 102.0 (5.18) | 101.6 (5.06)
SBPday [Mean (Standard Deviation); unit: mmHg] — Baseline SBPday [mean daytime (8 AM to 4 PM) ABPM SBP] was measured after the run-in period & prior to the 1st randomized dose (Day 3 to pre-dose Day 4). An Investigational Site member placed the cuff on the subject's non-dominant arm & connected the ABPM at approximately 7 AM (± 60 minutes) on Day 3. A pre-dose ABPM reading was recorded immediately prior to the morning dose of run-in period placebo (Day 3). The ABPM was started again immediately after dosing, and was removed at approximately 8 AM (± 60 minutes) on Day 4, but no sooner than 24 hours after the monitoring was initiated.
  mmHg | 149.8 (13.27) | 147.4 (9.61) | 149.1 (12.22)
SBPnight [Mean (Standard Deviation); unit: mmHg] — Baseline SBPnight [mean nighttime (10 PM to 6 AM) ABPM SBP] was measured after the run-in period & prior to the 1st randomized dose (Day 3 to pre-dose Day 4). An Investigational Site member placed the cuff on the subject's non-dominant arm & connected the ABPM at approximately 7 AM (± 60 minutes) on Day 3. A pre-dose ABPM reading was recorded immediately prior to the morning dose of run-in period placebo (Day 3). The ABPM was started again immediately after dosing, and was removed at approximately 8 AM (± 60 minutes) on Day 4, but no sooner than 24 hours after the monitoring was initiated.
  mmHg | 138.0 (17.34) | 133.3 (9.31) | 136.7 (15.48)
SBP24hr [Mean (Standard Deviation); unit: mmHg] — Baseline SBP24hr (mean 24-hour ABPM SBP) was measured after the run-in period & prior to the 1st randomized dose (Day 3 to pre-dose Day 4). An Investigational Site member placed the cuff on the subject's non-dominant arm & connected the ABPM at approximately 7 AM (± 60 minutes) on Day 3. A pre-dose ABPM reading was recorded immediately prior to the morning dose of run-in period placebo (Day 3). The ABPM was started again immediately after dosing, and was removed at approximately 8 AM (± 60 minutes) on Day 4, but no sooner than 24 hours after the monitoring was initiated.
  mmHg | 145.3 (14.02) | 141.2 (8.07) | 144.2 (12.62)
DBPday [Mean (Standard Deviation); unit: mmHg] — Baseline DBPday [mean daytime (8 AM to 4 PM) ABPM DBP] was measured after the run-in period & prior to the 1st randomized dose (Day 3 to pre-dose Day 4). An Investigational Site member placed the cuff on the subject's non-dominant arm & connected the ABPM at approximately 7 AM (± 60 minutes) on Day 3. A pre-dose ABPM reading was recorded immediately prior to the morning dose of run-in period placebo (Day 3). The ABPM was started again immediately after dosing, and was removed at approximately 8 AM (± 60 minutes) on Day 4, but no sooner than 24 hours after the monitoring was initiated.
  mmHg | 92.6 (11.20) | 93.3 (9.81) | 92.8 (10.61)
DBPnight [Mean (Standard Deviation); unit: mmHg] — Baseline DBPnight [mean nighttime (10 PM to 6 AM) ABPM DBP] was measured after the run-in period & prior to the 1st randomized dose (Day 3 to pre-dose Day 4). An Investigational Site member placed the cuff on the subject's non-dominant arm & connected the ABPM at approximately 7 AM (± 60 minutes) on Day 3. A pre-dose ABPM reading was recorded immediately prior to the morning dose of run-in period placebo (Day 3). The ABPM was started again immediately after dosing, and was removed at approximately 8 AM (± 60 minutes) on Day 4, but no sooner than 24 hours after the monitoring was initiated.
  mmHg | 82.3 (12.14) | 82.6 (3.23) | 82.4 (10.38)
DBP24hr [Mean (Standard Deviation); unit: mmHg] — Baseline DBP24hr (mean 24-hour ABPM DBP) was measured after the run-in period & prior to the 1st randomized dose (Day 3 to pre-dose Day 4). An Investigational Site member placed the cuff on the subject's non-dominant arm & connected the ABPM at approximately 7 AM (± 60 minutes) on Day 3. A pre-dose ABPM reading was recorded immediately prior to the morning dose of run-in period placebo (Day 3). The ABPM was started again immediately after dosing, and was removed at approximately 8 AM (± 60 minutes) on Day 4, but no sooner than 24 hours after the monitoring was initiated.
  mmHg | 88.6 (10.91) | 88.8 (6.04) | 88.7 (9.69)
Total Serum Magnesium AUC [Mean (Standard Deviation); unit: mEq*24hr/L] — Venous blood samples were collected within 1 hour prior to & 0.5, 1, 2, 3, 6, & 12 hours following the morning dose of run-in placebo on Day 3 & within 1 hour prior to the 1st randomized dose on Day 4. Blood samples were processed to serum & assayed for total serum magnesium by a central laboratory [lower limit of quantitation (LLOQ) = 0.06 mEq/L]. Individual concentration-time curves were plotted & area under the serum concentration-time curve from time zero to 24 hours post-dose (AUC0-24) values were derived. This value represents the subject's endogenous levels of total serum magnesium.
  mEq*24hr/L | 41.4 (2.42) | 42.8 (2.76) | 41.8 (2.53)
Total Serum Magnesium Concentration [Mean (Standard Deviation); unit: mEq/L] — A venous blood sample was collected within 1 hour prior to the first randomized dose (pre-dose Day 4). The blood sample was processed to serum & assayed for total serum magnesium by a central laboratory (LLOQ = 0.06 mEq/L). This value represents the subject's baseline concentration of endogenous total serum magnesium.
  mEq/L | 1.75 (0.103) | 1.78 (0.117) | 1.76 (0.105)
24-hour urinary magnesium excretion [Mean (Standard Deviation); unit: mEq/24 hrs] — Baseline urinary excretion of magnesium was assessed over a 24-hour period, starting immediately after the morning dose of run-in placebo on Day 3 and ending prior to the first randomized dose (i.e., Day 3 - pre-dose Day 4). This value represents the subject's baseline endogenous urinary magnesium excretion.
  mEq/24 hrs | 7.3 (2.59) | 7.0 (4.34) | 7.2 (3.05)
12-lead ECG Ventricular Rate [Mean (Standard Deviation); unit: bpm] — Baseline 12-lead electrocardiogram (ECG) ventricular rate was measured at Screening or Day 1. The ECG assessments were recorded after the subject was resting at least 5 minutes in the supine position in a quiet environment.
  bpm | 70.31 (9.904) | 65.83 (14.851) | 69.09 (11.258)
12-Lead ECG Intervals [Mean (Standard Deviation); unit: msec] — Baseline 12-lead ECG intervals (RR interval, PR interval, QRS interval, QT interval, corrected QT interval based on Fridericia formula) were measured at Screening or Day 1. The ECG assessments were recorded after the subject was resting at least 5 minutes in the supine position in a quiet environment.
  msec
    RR Interval | 863.31 (113.781) | 944.17 (199.272) | 885.36 (141.635)
    PR Interval | 168.38 (18.143) | 155.67 (10.985) | 164.91 (17.246)
    QRS Interval | 90.00 (9.033) | 97.67 (19.159) | 92.09 (12.566)
    QT Interval | 398.56 (24.916) | 416.00 (48.233) | 403.32 (32.566)
    Corrected QT Interval | 416.25 (21.592) | 424.00 (23.639) | 418.36 (21.875)
12-Lead ECG Diagnosis [Count of Participants; unit: Participants] — Baseline 12-lead ECG diagnosis [normal; abnormal but not clinically significant (NCS); abnormal and clinically significant (CS)] was assessed at Screening or Day 1. The ECG was recorded after the subject was resting at least 5 minutes in the supine position in a quiet environment.
  Participants
    Normal | 9 | 3 | 12
    Abnormal NCS | 7 | 3 | 10
    Abnormal CS | 0 | 0 | 0
Patellar Reflex Score [Count of Participants; unit: Participants] — Baseline patellar reflex score was measured at pre-dose Day 4. The scoring values included 0, 1+, 2+, 3+, and 4+, where 2+ means normal patellar reflex and lower scores indicate a worsened outcome (1+ means reflex present only with reinforcement and 0 means loss of reflex). The patellar reflex assessment was made with the subject in the seated position, with legs hanging freely from the exam table.
  Participants
    2+ | 11 | 6 | 17
    1+ | 5 | 0 | 5

OUTCOME MEASURES:

1. Primary Outcome: Safety and Tolerability of RMJH-111b Compared to Placebo Based on Treatment Emergent Adverse Events (TEAEs)
Description: Safety & tolerability were primarily assessed based on the incidence of reported TEAEs by system organ class & preferred term, as well as by categories: TEAE, severe TEAE, serious TEAE, drug-related TEAE, drug-related severe TEAE, drug-related serious TEAE, TEAE leading to discontinuation, & TEAE with outcome of death. Drug-related TEAEs were defined as TEAEs assigned a Study Drug (active or placebo) relationship of "adverse reaction" or "suspected adverse reaction".
  TEAEs were coded using the Medical Dictionary for Regulatory Activities, version 19.0. The severity of TEAEs were graded according to the National Cancer Institute Common Terminology Criteria for Adverse Events, version 4.03. TEAEs were defined as any adverse event that started or increased in severity after the first randomized dose of Study Drug on Day 4 through the Final Study Visit (8 +/-3 days after last randomized dose).
Time Frame: 14 days +/- 3 days
Population: Safety population = all randomized subjects who received at least one dose of Study Drug (active or placebo).
Measure: Count of Participants; unit: Participants
Arm/Group | RMJH-111b | Placebo
Number analyzed (Participants) | 16 | 6
Participants
  TEAE | 5 | 1
  Severe TEAE | 0 | 0
  Serious TEAE | 0 | 0
  Drug-related TEAE | 2 | 0
  Drug-related severe TEAE | 0 | 0
  Drug-related serious TEAE | 0 | 0
  TEAE leading to discontinuation from study | 0 | 0
  TEAE with outcome of death | 0 | 0
  Mild abdominal pain upper | 1 | 0
  Moderate constipation | 1 | 0
  Mild diarrhoea | 2 | 0
  Mild flatulence | 1 | 0
  Mild headache | 1 | 1
  Mild cough | 2 | 0

2. Primary Outcome: Safety and Tolerability of RMJH-111b Compared to Placebo Based on Change in 24-hour Urinary Magnesium Excretion
Description: Change in the mean value of 24-hour urinary magnesium excretion from baseline (Day 3 to pre-dose Day 4) to end of treatment (Day 10 to Day 11). Mean values that are negative represent a decrease in that value from baseline, whereas values that are positive represent an increase.
Time Frame: 8 days
Population: Safety population = all randomized subjects who received at least 1 dose of Study Drug. 1 subject in RMJH-111b arm was discontinued on Day 9 due to protocol-specified criterion [SBP<110 mmHg; the SBPs (102-109 mmHg) were not associated with clinical symptoms & were not assigned as TEAEs] & is therefore missing Day 10-11 assessment (i.e., n=15).
Measure: Mean (Standard Deviation); unit: mEq/24 hours
Arm/Group | RMJH-111b | Placebo
Number analyzed (Participants) | 15 | 6
mEq/24 hours | 9.1 (5.44) | -1.3 (5.57)

3. Primary Outcome: Safety and Tolerability of RMJH-111b Compared to Placebo Based on Change in Seated SBP and DBP
Description: Changes in the mean values for seated SBP & DBP from baseline (pre-dose Day 4) to end of treatment (Day 11). Mean values that are negative represent a decrease in that value from baseline, whereas values that are positive represent an increase.
Time Frame: 7 days
Population: Safety population = all randomized subjects who received at least 1 dose of Study Drug. 1 subject in RMJH-111b arm was discontinued on Day 9 due to protocol-specified criterion [SBP<110 mmHg; the SBPs (102-109 mmHg) were not associated with clinical symptoms & were not assigned as TEAEs] & is therefore missing Day 11 assessments (i.e., n=15).
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | RMJH-111b | Placebo
Number analyzed (Participants) | 15 | 6
mmHg
  Change in seated SBP | -14.6 (13.58) | -7.2 (7.36)
  Change in seated DBP | -6.4 (6.08) | -2.3 (6.25)

4. Primary Outcome: Safety and Tolerability of RMJH-111b Compared to Placebo Based on Change in Body Weight
Description: Change in mean body weight from baseline (Day 1) to end of treatment (Day 11). The weight measurements were made using a calibrated scale with the subject wearing light clothes and no shoes. Mean values that are negative represent a decrease in that value from baseline, whereas values that are positive represent an increase.
Time Frame: 10 days
Population: Safety population = all randomized subjects who received at least 1 dose of Study Drug. 1 subject in RMJH-111b arm was discontinued on Day 9 due to protocol-specified criterion [SBP<110 mmHg; the SBPs (102-109 mmHg) were not associated with clinical symptoms & were not assigned as TEAEs] & is therefore missing Day 11 assessment (i.e., n=15).
Measure: Mean (Standard Deviation); unit: kg
Arm/Group | RMJH-111b | Placebo
Number analyzed (Participants) | 15 | 6
kg | -1.09 (2.372) | -0.79 (1.421)

5. Primary Outcome: Safety and Tolerability of RMJH-111b Compared to Placebo Based on Change in 12-lead ECG Ventricular Rate (3 Hours After 1st Dose)
Description: Change in mean 12-lead ECG ventricular rate from baseline (Screening or Day 1) to 3 hours after the first randomized dose (Day 4). Mean values that are negative represent a decrease in that value from baseline, whereas values that are positive represent an increase. The ECG assessments were recorded after the subject was resting at least 5 minutes in the supine position in a quiet environment.
Time Frame: Up to 6 days
Population: Safety population = all randomized subjects who received at least 1 dose of Study Drug
Measure: Mean (Standard Deviation); unit: bpm
Arm/Group | RMJH-111b | Placebo
Number analyzed (Participants) | 16 | 6
bpm | -0.31 (8.554) | -5.17 (6.735)

6. Primary Outcome: Safety and Tolerability of RMJH-111b Compared to Placebo Based on Change in 12-lead ECG Ventricular Rate (After Last Dose)
Description: Change in mean 12-lead ECG ventricular rate from baseline (Screening or Day 1) to after the last randomized dose (Day 11). Mean values that are negative represent a decrease in that value from baseline, whereas values that are positive represent an increase. The ECG assessments were recorded after the subject was resting at least 5 minutes in the supine position in a quiet environment.
Time Frame: Up to 13 days
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: bpm
Arm/Group | RMJH-111b | Placebo
Number analyzed (Participants) | 15 | 6
bpm | 4.73 (10.579) | -3.83 (8.519)

7. Primary Outcome: Safety and Tolerability of RMJH-111b Compared to Placebo Based on Change in 12-lead ECG Intervals (3 Hours After 1st Dose)
Description: Change in mean 12-lead ECG intervals (RR interval, PR interval, QRS interval, QT interval, corrected QT interval based on Fridericia formula) from baseline (Screening or Day 1) to 3 hours after the first randomized dose (Day 4). Mean values that are negative represent a decrease in that value from baseline, whereas values that are positive represent an increase. The ECG assessments were recorded after the subject was resting at least 5 minutes in the supine position in a quiet environment.
Time Frame: Up to 6 days
Population: Safety population = all randomized subjects who received at least 1 dose of Study Drug
Measure: Mean (Standard Deviation); unit: msec
Arm/Group | RMJH-111b | Placebo
Number analyzed (Participants) | 16 | 6
msec
  Change in RR Interval | 8.06 (102.179) | 55.33 (96.804)
  Change in PR Interval | 0.75 (13.364) | 8.67 (4.502)
  Change in QRS Interval | -2.63 (4.113) | 2.33 (4.274)
  Change in QT Interval | -5.06 (26.727) | -0.33 (23.372)
  Change in Corrected QT Interval | -5.06 (16.097) | -9.17 (16.005)

8. Primary Outcome: Safety and Tolerability of RMJH-111b Compared to Placebo Based on Change in 12-lead ECG Intervals (After Last Dose)
Description: Change in mean 12-lead ECG intervals (RR interval, PR interval, QRS interval, QT interval, corrected QT interval based on Fridericia formula) from baseline (Screening or Day 1) to after the last randomized dose (Day 11). Mean values that are negative represent a decrease in that value from baseline, whereas values that are positive represent an increase. The ECG assessments were recorded after the subject was resting at least 5 minutes in the supine position in a quiet environment.
Time Frame: Up to 13 days
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: msec
Arm/Group | RMJH-111b | Placebo
Number analyzed (Participants) | 15 | 6
msec
  Change in RR Interval | -57.00 (122.412) | 29.67 (82.921)
  Change in PR Interval | -4.00 (12.806) | 8.33 (13.530)
  Change in QRS Interval | -1.33 (3.677) | -0.67 (5.317)
  Change in QT Interval | -11.67 (24.732) | 5.67 (22.393)
  Change in Corrected QT Interval | -1.47 (11.332) | -0.33 (12.307)

9. Primary Outcome: Safety and Tolerability of RMJH-111b Compared to Placebo Based on Change in 12-lead ECG Diagnosis (3 Hours After 1st Dose)
Description: Change in 12-lead ECG diagnosis [i.e., normal to abnormal not clinically significant (NCS); normal to abnormal clinically significant (CS); abnormal NCS to abnormal CS; remained abnormal NCS; remained normal] from baseline (Screening or Day 1) to 3 hours after the first randomized dose (Day 4). The ECG was recorded after the subject was resting at least 5 minutes in the supine position in a quiet environment.
Time Frame: Up to 6 days
Population: Safety population = all randomized subjects who received at least 1 dose of Study Drug
Measure: Count of Participants; unit: Participants
Arm/Group | RMJH-111b | Placebo
Number analyzed (Participants) | 16 | 6
Participants
  Changed from Normal to Abnormal NCS | 1 | 1
  Changed from Normal to Abnormal CS | 0 | 0
  Changed from Abnormal NCS to Abnormal CS | 0 | 0
  Remained Abnormal NCS | 7 | 3
  Remained Normal | 8 | 2

10. Primary Outcome: Safety and Tolerability of RMJH-111b Compared to Placebo Based on Change in 12-lead ECG Diagnosis (After Last Dose)
Description: Change in 12-lead ECG diagnosis [i.e., normal to abnormal not clinically significant (NCS); normal to abnormal clinically significant (CS); abnormal NCS to abnormal CS; remained abnormal NCS; remained normal] from baseline (Screening or Day 1) to after the last randomized dose (Day 11). The ECG was recorded after the subject was resting at least 5 minutes in the supine position in a quiet environment.
Time Frame: Up to 13 days
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | RMJH-111b | Placebo
Number analyzed (Participants) | 15 | 6
Participants
  Changed from Normal to Abnormal NCS | 1 | 0
  Changed from Normal to Abnormal CS | 0 | 0
  Changed from Abnormal NCS to Abnormal CS | 0 | 0
  Remained Abnormal NCS | 6 | 2
  Remained Normal | 7 | 3
  Changed from Abnormal NCS to Normal | 1 | 1

11. Primary Outcome: Safety and Tolerability of RMJH-111b Compared to Placebo Based on Change in Patellar Reflex Score
Description: Changes in patellar reflex score from baseline (pre-dose Day 4) to interim time points during the randomized treatment period (prior to each morning dose on Days 5 through 10) and to post-dose time points (Day 11 & Day 18 ± 3 days). The scoring values included 0, 1+, 2+, 3+, and 4+, where 2+ means normal patellar reflex and lower scores indicate a worsened outcome (1+ means reflex present only with reinforcement and 0 means loss of reflex). The patellar reflex assessment was made with the subject in the seated position, with legs hanging freely from the exam table.
  Loss of patellar reflex is an early sign of magnesium toxicity, and thus the test serves as an assessment for functional magnesium status. A clinical indication of a safe magnesium dosage regimen included the presence of the patellar reflex (knee jerk).
Time Frame: 14 days +/- 3 days
Population: Safety population = all randomized subjects who received at least 1 dose of Study Drug. 1 RMJH-111b subject was discontinued on Day 9 due to protocol requirement [SBP<110 mmHg; SBPs (102-109 mmHg) not associated with clinical symptoms & not assigned as TEAEs] & lacked Day 10-11 assessments (i.e., n=15). Subject was at 2+ for Day 4-9 & Final Visit.
Measure: Count of Participants; unit: Participants
Arm/Group | RMJH-111b | Placebo
Number analyzed (Participants) | 15 | 6
Participants
  Remained at 2+ | 9 | 6
  Remained at 1+ | 2 | 0
  Remained at 2+ except Day 9 (1+) | 1 | 0
  Remained at 1+ except Day 5 & 8 (2+) | 1 | 0
  Remained at 1+ except Day 18 (2+) | 1 | 0
  Remained 1+ except Days 6, 10, & 11 (2+) | 1 | 0

12. Secondary Outcome: Pharmacokinetics of Total Serum Magnesium After Single and Repeated Oral Administrations of RMJH-111b Compared to Placebo Based on AUC
Description: Venous blood samples were collected within 1 hour prior to & 0.5, 1, 2, 3, 6, & 12 hours following the morning dose of Study Drug on Days 3 (run-in placebo) and 4, & within 1 hour prior to & 0.5, 1, 2, 3, 6, 12, & 24 hours following the morning dose of Study Drug on Day 10. Blood samples were processed to serum & assayed for total serum magnesium by a central laboratory. The LLOQ was 0.06 mEq/L.
  Individual PK parameters for Days 4 & 10 were to be calculated using corrected concentration-time curves (with individual's baseline assessments of endogenous total serum magnesium at Day 3 subtracted); however, due to small numerical values after correction, the planned PK parameters could not be derived. The analyses were reattempted using the observed values (that include the endogenous levels of magnesium), which allowed AUC0-24 to be derived.
Time Frame: 8 days
Population: PK population = all randomized subjects who received at least 1 dose of Study Drug with valid data for at least 1 pre- & post-dose assessment. 1 subject in RMJH-111b arm was missing PK assessments beyond Day 8, & thus is only included in the analyses for Days 3 & 4 and not for Day 10 (i.e., n = 16 for Days 3 & 4, but n = 15 for Day 10).
Measure: Mean (Standard Deviation); unit: mEq*24hr/L
Arm/Group | RMJH-111b | Placebo
Number analyzed (Participants) | 16 | 6
mEq*24hr/L
  Day 3 (pre-dose) | 41.4 (2.42) | 42.8 (2.76)
  Day 4 (1st day of dosing) | 43.9 (2.53) | 42.4 (3.03)
  Day 10 (7th day of dosing) | 43.9 (1.87) | 41.7 (2.52)

13. Secondary Outcome: Pharmacokinetics of Total Serum Magnesium After Single and Repeated Oral Administrations of RMJH-111b Compared to Placebo Based on Trough Concentration Ratio
Description: Venous blood samples were collected within 1 hour prior to the morning dose of Study Drug (active or placebo) on Days 4, 5, 6, 7, 8, 9, and 10. Blood samples were processed to serum & assayed for total serum magnesium by a central laboratory (LLOQ = 0.06 mEq/L).
  Ratios of the individual total serum magnesium trough concentrations at Days 5, 6, 7, 8, 9, and 10 relative to baseline (pre-dose Day 4) were calculated. Observed concentrations (including the endogenous levels of magnesium) were used for this purpose.
Time Frame: 6 days
Population: PK population = all randomized subjects who received at least 1 dose of Study Drug with valid data for at least 1 pre- & post-dose assessment. 1 subject in RMJH-111b arm was missing PK assessments beyond Day 8, & thus is only included in the analyses for Days 5-8 and not for Days 9-10 (i.e., n = 16 for Days 5-8, but n = 15 for Days 9-10).
Measure: Mean (Standard Deviation); unit: unitless (i.e., ratio of mEq/L to mEq/L)
Arm/Group | RMJH-111b | Placebo
Number analyzed (Participants) | 16 | 6
unitless (i.e., ratio of mEq/L to mEq/L)
  Day 5/Day 4 trough concentrations | 1.09 (0.059) | 1.00 (0.034)
  Day 6/Day 4 trough concentrations | 1.10 (0.071) | 0.99 (0.041)
  Day 7/Day 4 trough concentrations | 1.08 (0.097) | 0.98 (0.045)
  Day 8/Day 4 trough concentrations | 1.09 (0.087) | 1.01 (0.043)
  Day 9/Day 4 trough concentrations | 1.06 (0.063) | 1.02 (0.058)
  Day 10/Day 4 trough concentrations | 1.02 (0.080) | 0.96 (0.028)

14. Secondary Outcome: Pharmacokinetics of Urine Magnesium After Single and Repeated Oral Administrations of RMJH-111b Compared to Placebo Based on 24-hour Urinary Excretion
Description: Urinary excretion of magnesium was assessed over three 24-hour periods. The first urine collection started immediately after the morning dose of run-in placebo on Day 3, and the second and third collections started immediately after the morning dose of Study Drug on Days 4 and 10, respectively.
  Observed 24-hour urinary magnesium excretion values at Days 3, 4, and 10 (i.e., without subtraction of the Day 3 values to correct for the individual's baseline assessment of endogenous urinary magnesium excretion) were used for comparisons with the total serum magnesium data (as only the observed serum values allowed for PK parameter derivation).
Time Frame: 8 days
Population: PK population = all randomized subjects who received at least 1 dose of Study Drug with valid data for at least 1 pre- & post-dose assessment. 1 subject in RMJH-111b arm was missing PK assessments beyond Day 8, & thus is only included in the analyses for Days 3 & 4 and not for Day 10 (i.e., n = 16 for Days 3 and 4, but n = 15 for Day 10).
Measure: Mean (Standard Deviation); unit: mEq/24 hrs
Arm/Group | RMJH-111b | Placebo
Number analyzed (Participants) | 16 | 6
mEq/24 hrs
  Day 3 (pre-dose) | 7.3 (2.59) | 7.0 (4.34)
  Day 4 (1st day of dosing) | 9.8 (3.90) | 5.7 (1.97)
  Day 10 (7th day of dosing) | 16.5 (6.23) | 5.7 (1.63)

15. Secondary Outcome: Efficacy of RMJH-111b Compared to Placebo Based on Change From Baseline in SBPday After 7 Days of Treatment
Description: SBPday = mean daytime (8 AM to 4 PM) ABPM SBP. Note, mean values of change that are negative represent a decrease in that value from baseline, whereas values that are positive represent an increase.
  SBPday was measured twice during the subject's stay at the CRU: baseline measurements were collected from Day 3 to pre-dose Day 4 & post-dose measurements were collected from Day 10 to Day 11. An Investigational Site staff member placed the cuff on the subject's non-dominant arm & connected the ABPM at approximately 7 AM (± 60 minutes) on Days 3 & 10. A pre-dose ABPM reading was recorded immediately prior to the morning dose of run-in period placebo on Day 3 & the morning dose of treatment period Study Drug (active or placebo) on Day 10. The ABPM was started again immediately after dosing. The ABPM was removed at approximately 8 AM (± 60 minutes) on Days 4 and 11, respectively, but no sooner than 24 hours after the continuous monitoring was initiated.
Time Frame: 8 days
Population: Efficacy population = all randomized subjects who completed 7 days of treatment & the Day 3-Day 4 and Day 10-Day 11 ABPM assessments. 1 subject in RMJH-111b arm was discontinued on Day 9 due to meeting protocol-specified criterion (SBP < 110 mmHg). The SBPs (102-109 mmHg) were not associated with clinical symptoms & were not assigned as TEAEs.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | RMJH-111b | Placebo
Number analyzed (Participants) | 15 | 6
mmHg | -4.6 (11.72) | 1.6 (11.36)

16. Secondary Outcome: Efficacy of RMJH-111b Compared to Placebo Based on Change From Baseline in SBPnight After 7 Days of Treatment
Description: SBPnight = mean daytime (10 PM to 6 AM) ABPM SBP. Note, mean values of change that are negative represent a decrease in that value from baseline, whereas values that are positive represent an increase.
  SBPnight was measured twice during the subject's stay at the CRU: baseline measurements were collected from Day 3 to pre-dose Day 4 & post-dose measurements were collected from Day 10 to Day 11. An Investigational Site staff member placed the cuff on the subject's non-dominant arm & connected the ABPM at approximately 7 AM (± 60 minutes) on Days 3 & 10. A pre-dose ABPM reading was recorded immediately prior to the morning dose of run-in period placebo on Day 3 & the morning dose of treatment period Study Drug (active or placebo) on Day 10. The ABPM was started again immediately after dosing. The ABPM was removed at approximately 8 AM (± 60 minutes) on Days 4 and 11, respectively, but no sooner than 24 hours after the continuous monitoring was initiated.
Time Frame: 8 days
Population: as for outcome 15
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | RMJH-111b | Placebo
Number analyzed (Participants) | 15 | 6
mmHg | -4.2 (12.54) | 0.7 (12.13)

17. Secondary Outcome: Efficacy of RMJH-111b Compared to Placebo Based on Change From Baseline in SBP24hr After 7 Days of Treatment
Description: SBP24hr = mean 24-hour ABPM SBP. Note, mean values of change that are negative represent a decrease in that value from baseline, whereas values that are positive represent an increase.
  SBP24hr was measured twice during the subject's stay at the CRU: baseline measurements were collected from Day 3 to pre-dose Day 4 & post-dose measurements were collected from Day 10 to Day 11. An Investigational Site staff member placed the cuff on the subject's non-dominant arm & connected the ABPM at approximately 7 AM (± 60 minutes) on Days 3 & 10. A pre-dose ABPM reading was recorded immediately prior to the morning dose of run-in period placebo on Day 3 & the morning dose of treatment period Study Drug (active or placebo) on Day 10. The ABPM was started again immediately after dosing. The ABPM was removed at approximately 8 AM (± 60 minutes) on Days 4 and 11, respectively, but no sooner than 24 hours after the continuous monitoring was initiated.
Time Frame: 8 days
Population: as for outcome 15
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | RMJH-111b | Placebo
Number analyzed (Participants) | 15 | 6
mmHg | -3.8 (11.72) | 2.3 (11.61)

18. Secondary Outcome: Efficacy of RMJH-111b Compared to Placebo Based on Change From Baseline in DBPday After 7 Days of Treatment
Description: DBPday = mean daytime (8 AM to 4 PM) ABPM DBP. Note, mean values of change that are negative represent a decrease in that value from baseline, whereas values that are positive represent an increase.
  DBPday was measured twice during the subject's stay at the CRU: baseline measurements were collected from Day 3 to pre-dose Day 4 & post-dose measurements were collected from Day 10 to Day 11. An Investigational Site staff member placed the cuff on the subject's non-dominant arm & connected the ABPM at approximately 7 AM (± 60 minutes) on Days 3 & 10. A pre-dose ABPM reading was recorded immediately prior to the morning dose of run-in period placebo on Day 3 & the morning dose of treatment period Study Drug (active or placebo) on Day 10. The ABPM was started again immediately after dosing. The ABPM was removed at approximately 8 AM (± 60 minutes) on Days 4 and 11, respectively, but no sooner than 24 hours after the continuous monitoring was initiated.
Time Frame: 8 days
Population: as for outcome 15
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | RMJH-111b | Placebo
Number analyzed (Participants) | 15 | 6
mmHg | -3.5 (6.88) | -1.2 (7.12)

19. Secondary Outcome: Efficacy of RMJH-111b Compared to Placebo Based on Change From Baseline in DBPnight After 7 Days of Treatment
Description: DBPnight = mean nighttime (10 PM to 6 AM) ABPM DBP. Note, mean values of change that are negative represent a decrease in that value from baseline, whereas values that are positive represent an increase.
  DBPnight was measured twice during the subject's stay at the CRU: baseline measurements were collected from Day 3 to pre-dose Day 4 & post-dose measurements were collected from Day 10 to Day 11. An Investigational Site staff member placed the cuff on the subject's non-dominant arm & connected the ABPM at approximately 7 AM (± 60 minutes) on Days 3 & 10. A pre-dose ABPM reading was recorded immediately prior to the morning dose of run-in period placebo on Day 3 & the morning dose of treatment period Study Drug (active or placebo) on Day 10. The ABPM was started again immediately after dosing. The ABPM was removed at approximately 8 AM (± 60 minutes) on Days 4 and 11, respectively, but no sooner than 24 hours after the continuous monitoring was initiated.
Time Frame: 8 days
Population: as for outcome 15
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | RMJH-111b | Placebo
Number analyzed (Participants) | 15 | 6
mmHg | -1.9 (8.76) | -0.6 (7.46)

20. Secondary Outcome: Efficacy of RMJH-111b Compared to Placebo Based on Change From Baseline in DBP24hr After 7 Days of Treatment
Description: DBP24hr = mean 24-hour ABPM DBP. Note, mean values of change that are negative represent a decrease in that value from baseline, whereas values that are positive represent an increase.
  DBP24hr was measured twice during the subject's stay at the CRU: baseline measurements were collected from Day 3 to pre-dose Day 4 & post-dose measurements were collected from Day 10 to Day 11. An Investigational Site staff member placed the cuff on the subject's non-dominant arm & connected the ABPM at approximately 7 AM (± 60 minutes) on Days 3 & 10. A pre-dose ABPM reading was recorded immediately prior to the morning dose of run-in period placebo on Day 3 & the morning dose of treatment period Study Drug (active or placebo) on Day 10. The ABPM was started again immediately after dosing. The ABPM was removed at approximately 8 AM (± 60 minutes) on Days 4 and 11, respectively, but no sooner than 24 hours after the continuous monitoring was initiated.
Time Frame: 8 days
Population: as for outcome 15
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | RMJH-111b | Placebo
Number analyzed (Participants) | 15 | 6
mmHg | -2.3 (6.97) | 0.3 (6.53)

21. Secondary Outcome: Efficacy of RMJH-111b Compared to Placebo Based on Change From Baseline in Seated SBP After 7 Days of Treatment
Description: Change from baseline (pre-dose Day 4) in seated SBP after 7 days of treatment (Day 11) with RMJH-111b compared to placebo was a secondary efficacy variable (i.e., seated SBP served dual functions as safety and efficacy variables, with the safety population used for the safety analyses described in outcome 3 and the efficacy population used for the efficacy analyses described here). Note, mean values that are negative represent a decrease in that value from baseline, whereas values that are positive represent an increase.
Time Frame: 7 days
Population: Efficacy population = all randomized subjects who completed 7 days of treatment & pre-dose Day 4 & Day 11 assessments. 1 subject in RMJH-111b arm was discontinued on Day 9 for meeting protocol-specified criterion [SBP<110 mmHg; SBPs (102-109 mmHg) were not associated with clinical symptoms & not assigned as TEAEs] & is therefore excluded.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | RMJH-111b | Placebo
Number analyzed (Participants) | 15 | 6
mmHg | -14.6 (13.58) | -7.2 (7.36)

22. Secondary Outcome: Efficacy of RMJH-111b Compared to Placebo Based on Change From Baseline in Seated DBP After 7 Days of Treatment
Description: Change from baseline (pre-dose Day 4) in seated DBP after 7 days of treatment (Day 11) with RMJH-111b compared to placebo was a secondary efficacy variable (i.e., seated DBP served dual functions as safety and efficacy variables, with the safety population used for the safety analyses described in outcome 3 and the efficacy population used for the efficacy analyses described here). Note, mean values that are negative represent a decrease in that value from baseline, whereas values that are positive represent an increase.
Time Frame: 7 days
Population: as for outcome 21
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | RMJH-111b | Placebo
Number analyzed (Participants) | 15 | 6
mmHg | -6.4 (6.08) | -2.3 (6.25)

ADVERSE EVENTS:
Time Frame: 14 +/- 3 days. Treatment emergent adverse events (TEAEs) were defined as any adverse event (AE) that started or increased in severity after the first randomized dose of Study Drug (active or placebo) on Day 4 through the Final Study Visit (8 +/-3 days after last randomized dose).
Description: AE = any untoward medical occurrence associated with use of Study Drug (active or placebo), whether or not considered drug related. Includes any unfavorable & unintended sign (e.g., an abnormal laboratory finding), symptom, or disease temporally associated with the use of the drug, & does not imply any judgment about causality. Can arise with any use of the drug (e.g., off-label use, use in combination with another drug) & any route of administration, formulation, or dose, including overdose.
Arm/Group | RMJH-111b | Placebo
All-Cause Mortality (participants affected / at risk) | 0/16 | 0/6
Serious Adverse Events (participants affected / at risk) | 0/16 | 0/6
Other Adverse Events (participants affected / at risk) | 5/16 | 1/6
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | RMJH-111b (N=16) | Placebo (N=6)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1) | 0 (0) — intermittent mild
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0) — continuous moderate
Diarrhoea (Gastrointestinal disorders) | 2 (2) | 0 (0) — single event or intermittent mild
Flatulence (Gastrointestinal disorders) | 1 (1) | 0 (0) — intermittent mild
Headache (Nervous system disorders) | 1 (1) | 1 (2) — intermittent mild
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) — intermittent mild

LIMITATIONS AND CAVEATS:
See Detailed Description under Study Description section of record for study design rationale and limits with regards to PK analysis of serum magnesium.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes